CLINICAL TRIAL: NCT01291290
Title: Thrombocyte Administration Versus no Thrombocytes to Patients With Ruptured Abdominal Aortic Aneurism Before Transport to Hospital With Vascular Surgical Department
Brief Title: START - Early Thrombocyte Administration to Patients With Ruptured Abdominal Aortic Aneurism
Acronym: rAAA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Thomas Bech Jorgensen, Afdelingslaege, Rigshospitalet, Denmark
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Treatment
Other Study IDs: H-D-2009-002
Record Dates: First submitted 2011-02-07; First posted 2011-02-08 (Estimated); Last update posted 2013-03-14 (Estimated); Status verified 2013-03

CONDITIONS: Ruptured Abdominal Aortic Aneurism
Keywords: rAAA; Platelets; TEG; Massive bleeding; Coagulopathy
MeSH Terms: conditions — Hemostatic Disorders | interventions — Platelet Count

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control treatment (No Intervention): Usual transfusion regime to patients with rAAA
- Thrombocyte (Experimental): Early thrombocyte administration to patients with rAAA
  Interventions: Procedure: Platelet

INTERVENTIONS:
Procedure: Platelet — 2 portions of platelets (one portion = pooled from 4 donors, 350ml) infused when diagnosed with rAAA and vascular surgeon accepts to receive the patient, infused before transportation.
  Other Names: Thrombocyte; Platelets
  Arms: Thrombocyte

SUMMARY:
The purpose of this study is to investigate the effect of platelet infusion prior to transfer to a vascular surgical department in patients with a ruptured abdominal aortic aneurism.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed with rAAA either by clinical evaluation or CT or UL

Exclusion Criteria:

* formerly randomized in the study
* aneurism not ruptured during operation

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 420 (Estimated)
Dates: Start 2010-03; Primary Completion 2014-03 (Estimated); Study Completion 2015-03 (Estimated)

PRIMARY OUTCOMES:
Mortality | 30 days
  Mortality during the first 30days after randomization, and time to death during the 30 days.

SECONDARY OUTCOMES:
Acute myocardial infarction | 30 days
  Development of AMI during the first 30 days after randomization, and the time to development during the first 30 days.
Post operative kidney failure | 30 days
  The need for dialysis during the first 30 days, time to start of dialysis and length.
Post operative pulmonary insufficiency | 30 days
  Length of respirator treatment in the ICU during the first 30 days.
Length of stay in ICU | until discharged from ICU
  Length of stay in ICU
Length of stay in hospital | until discharged from hospital
  Until discharged from main surgical department or if transferred to local hospital, when the patient leave local hospital.

CONTACTS AND LOCATIONS:
Overall Officials: Henning Bay Nielsen, MD, Study Chair
Locations (1):
- Rigshospitalet, Copenhagen, Oesterbro, Denmark